CLINICAL TRIAL: NCT06398353
Title: Investigating the Impact of Acupuncture on the Quality of Life of Primitive Headaches Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 232
Record Dates: First submitted 2024-03-18; First posted 2024-05-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-01

CONDITIONS: Headache Migraine
Keywords: Headache; Migraine
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture (Experimental)
  Interventions: Other: Real acupuncture; Other: Sham acupuncture
- sham acupuncture (Sham Comparator)
  Interventions: Other: Real acupuncture; Other: Sham acupuncture

INTERVENTIONS:
Other: Real acupuncture — Real acupuncture twice a week for two weeks
Other: Sham acupuncture — Sham acupuncture twice a week for two weeks

SUMMARY:
Primary headache is one of the most common neurological diseases in modern society, which seriously affects the patient's quality of life. Although the use of painkillers can alleviate primary headache symptoms, it may also cause drug dependence. Therefore, alternative therapies that do not rely on drugs have attracted increasing attention in recent years. Among them, acupuncture has been partially recognized by the public as an effective treatment for primary headaches. However, there is currently no scientific evidence that acupuncture is effective for primary headaches. The purpose of this project is to verify the effect of acupuncture in treating primary headaches. This study has three sub-projects:

Subproject 2 explores the impact of acupuncture on headache severity and quality of life in patients with primary headaches. We evaluate the quality of life before and after acupuncture treatment through professional questionnaires, including the Numerical rating scale (NRS), headache diary, depression, anxiety and stress scale (DASS-21), health quality of life measurement questionnaire, Migraine Disability Assessment Scale and SF-36 Taiwan version. Finally, these data will be combined with the pulseway analysis from the results of sub-project 1 to provide a comprehensive way to evaluate the treatment effect.

DETAILED DESCRIPTION:
In this study, 120 subjects who already suffered from headache symptoms (such as dizziness, heavy head, lightheadedness, head fullness, migraine) were treated with acupuncture at acupuncture points, and the pulse diagnosis instrument was used to capture the subjects' symptoms during acupuncture. The pulse waves before and after are collected, compared and analyzed to complete this test.

After the subjects are accepted, they will go to the Acupuncture and Traumatology Department of the Department of Traditional Chinese Medicine of Chang Gung Memorial Hospital (Taoyuan Branch) at an agreed time for health education and filling out questionnaires. After filling out the questionnaire, participants can reserve a time for the test.

One person is tested each time, and each test lasts 70-80 minutes. Pulse waves are collected for 20 minutes before and after the test. The acupuncture treatment plan for each subject in this study was based on traditional Chinese medicine theory and published literature. The acupuncture points selected were bilateral Cuanzhu, Taiyang, Tianzhu, Fengchi, Baihui, Hegu, Neiting, Zusanli, Waiguan, and Zulin. Qi, Houxi, Shenmai, Taichong. The doctor will select the above 4-6 acupoints according to the disease. It is divided into an acupuncture group and a sham acupuncture group. Before the experiment, first fill out the questionnaire. This trial is divided into an acupuncture group and a sham acupuncture group. A crossover design is adopted. 50% of the subjects will be assigned to the acupuncture group first. Then they will be connected to the sham acupuncture group, and the other 50% of the subjects will be assigned to the sham acupuncture group first and then the acupuncture group. Each group will last for two weeks, and acupuncture will be performed twice a week at the set acupuncture points. The first group of acupuncture will end. , will be interrupted for two weeks, and then another set of tests will be conducted, and then the patient will go to Chang Gung Memorial Hospital Taoyuan Branch for the final scale and quality of life questionnaire. The total trial period was eight weeks.

While undergoing the test, try to avoid taking Chinese and Western medicines and alcoholic beverages to avoid interfering with the study. (If participants usually take antihypertensive drugs and heart drugs, participants can continue to take them.) After the test, participants should drink more warm water and get enough rest. Do not take a shower or touch or drink cold things.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign a written subject consent form
2. Male or female over 18 years old
3. Those who have headaches (for example: dizziness, heavy head, dizziness, head fullness, migraine), those who have headaches more than twice a week, and whose NRS score is ˃ 4.
4. Headache definition: Headache symptoms are classified according to the ICHD-3 headache classification of the International Headache Organization, and are mainly primary headaches.

Dr. Chang ,Y.-J. and Dr. Yang ,C.-C. help to exclude headache patients with the following exclusion conditions to reduce the risk to subjects.

Exclusin Criteria

1. Pregnant women
2. Various acute and chronic infectious diseases, various skin ulcers, sores, burns, etc.
3. The patient has injuries to the radial artery or wrist, or has steel nails, plates, or fractures.
4. Various types of headaches related to anatomical structural lesions
5. Headaches associated with taking or withdrawing from substances (drugs, food, or other chemicals)
6. Headaches related to non-head infections and metabolic diseases
7. People with painful cranial neuropathy, other facial pain and other headaches
8. People with secondary headaches according to ICHD-3 beta
9. Other patients who have been evaluated by physicians as not suitable for inclusion in the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | 2 minutes
  Numerical rating scale (NRS) is the most commonly used pain intensity assessment tool at home and abroad. A straight line that is actually 10 centimeters, marked with "0" on the far left and "10" on the far right. Explain to the patient that "0" means no pain and "10" means very painful. The pain level increases from left to right, so that the patient can Draw vertically with a pen a few centimeters where the pain feels and record it in centimeters. You can also simply explain to the patient orally the meaning represented by "0" to "10" and let the patient rate it (verbal rating).
The Depression, Anxiety and Stress Scale (DASS-21), | 7minutes
  The Depression, Anxiety and Stress Scale (DASS-21), also known as the "Self-Rating Emotion Scale" is a self-report scale that effectively assesses depression, anxiety and stress levels of the general population; it has 21 questions in total and takes time About 5 minutes. Although this scale cannot replace professional clinical diagnosis, nor can it be used as a basis for diagnosis alone, it has a significant screening effect on minor mental health problems.
Europe health-related quality of life questionnaire 5 dimensions (EQ-5D) | 7minutes
  Europe health-related quality of life questionnaire 5 dimensions (EQ-5D) is a preference-based health life quality measurement tool. It includes 5 self-classifier questions and 0 - Two parts including a 100-point self-assessment scale for current health status.
The headache diary | 20minutes
  The headache diary is to record your own headache diary every day, which can make it easier to communicate with the doctor about your pain condition and help the doctor treat primary headaches.
Migraine Disability Assessment Questionnaire (MIDAs) | 7minutes
  Migraine Disability Assessment Questionnaire (MIDAs) In 1999, Stewart and Lipton proposed the Migraine Disability Assessment Questionnaire (MIDAs). This scale mainly consists of five questions, asking the patient to recall the impact of migraine on schoolwork or work, household affairs, and family, social or leisure activities during the past three months. This questionnaire is also used in Japan, Upper Turkey, Italy and other countries because it is simple and easy to use and has good reliability, validity and objectivity evaluation.
The Taiwan Short Form 36 Health Scale (SF-36) | 20minutes
  The Taiwan Short Form 36 Health Scale (SF-36) is a widely used health-related quality of life questionnaire and is also used by people with different cultural backgrounds. Research results show that SF36 has been proven to have good reliability and validity regardless of the diagnosis, age, and gender of the test subjects, and it can also sensitively detect changes before and after treatment without falling. Therefore, this study uses SF36 as the outcome measurement tool for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung YANG, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Select A State, Taiwan

IPD SHARING:
Plan to Share IPD: No